CLINICAL TRIAL: NCT06156215
Title: PROmotion of COVID-19 BOOSTer VA(X)Ccination in the Emergency Department - PROBOOSTVAXED
Acronym: PROBOOSTVAXED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Pfizer (Industry); Duke University (Other); Baylor College of Medicine (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 23-39854; R01AI166967-01 (NIH)
Record Dates: First submitted 2023-12-01; First posted 2023-12-05 (Actual); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: COVID-19
Keywords: COVID-19; health disparities; booster vaccines; healthcare access; vaccination; public health
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: PROBOOSTVAXED has 3 arms:
  Intervention M (Messaging + Vaccine Question)
  * Vaccine messaging given
  * Vaccine acceptance question asked
  Intervention Q (Vaccine Question, No Messaging)
  * No vaccine messaging
  * Vaccine acceptance question asked
  Control (No Messaging, No Vaccine Question)
  * No vaccine messaging
  * No vaccine acceptance question
Who Masked: Outcomes Assessor
Masking Description: Outcomes will be assessed at 30 days via EHR review or follow up phone call. EHR review and follow up calls will be conducted in a blinded fashion - the research staff person reviewing outcomes will be unaware of participant's study group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) (Experimental): * Vaccine messaging
  * Vaccine acceptance question All patients will receive an Intake Survey assessing their demographic and vaccination information.
  At the end of the Intake Survey, the Clinical Research Coordinator (CRC) will deliver the booster vaccine information flyer and ask the patient if they will watch a short video on booster vaccines. If they agree, the CRC will give them a QR code to view the video on their smartphone or an iPad. After finishing with the video, the CRC will tell the subject that they will be back for the Vaccine Acceptance survey. The CRC will then leave the room and ask the patient's primary provider to deliver the booster vaccine scripted message. This message is short and should not significantly impact provider workflow.
  Vaccine Acceptance Survey (Post-Intervention) in the ED: We will administer the Vaccine Acceptance Survey at 30 minutes to 3 hours after the Intake Survey.
  Interventions: Behavioral: Vaccine Messaging; Behavioral: Vaccine Acceptance Question
- Intervention Q (Vaccine Question, No Messaging) (Active Comparator): * No vaccine messaging
  * Vaccine acceptance question asked in the Vaccine Acceptance Survey
  Vaccine Acceptance Survey: We will administer the Vaccine Acceptance Survey at some time (generally 30 minutes but up to 3 hours) after the Intake Survey. The surveys in the control group retain the same key primary and secondary outcome questions as in the intervention group Vaccine Acceptance surveys.
  Interventions: Behavioral: Vaccine Acceptance Question
- Control (No Messaging, No Vaccine Question) (No Intervention): * No vaccine messaging
  * No vaccine acceptance question
  The workflow during this arm is identical to the Intervention Q arm except there will be no Vaccine Acceptance Question survey.

INTERVENTIONS:
Behavioral: Vaccine Messaging — 1. Video clips - short (approximately 3-minute) Public Service Announcement type videos to be viewed by participant using a QR code on their smartphone. If no smartphone is available, the video will be shown to the participant on an iPad.
  2. Printed materials - one page information sheets handed to subjects by CRCs.
  3. Face to face messaging - short (< 1 minute), scripted message from the patient's providers in the ED (nurse or provider)
  Each site will maintain a library of
  A. 5 versions of the videos - the version used in any participant will be tailored to that participant's stated race/ethnicity.
  B. 5 versions of printed flyers - likewise, the version will be tailored to the participant's stated race/ethnicity.
  C. 1 version of scripted message to be delivered in English or Spanish.
  Arms: PROBOOSTVAXED Intervention M (Messaging + Vaccine Question)
Behavioral: Vaccine Acceptance Question — The last question in the Vaccine Acceptance Survey in both the Intervention M and Intervention Q arms of the study is "Would you accept the COVID-19 booster vaccine in the emergency department today if your doctor asked you?"
  Arms: Intervention Q (Vaccine Question, No Messaging); PROBOOSTVAXED Intervention M (Messaging + Vaccine Question)

SUMMARY:
The goal of this cluster randomized clinical trial is to test the efficacy of messaging interventions to increase booster vaccine uptake in adults in the emergency department(ED). The main question[s] and goals of this study are:

* does the intervention of vaccine messaging increase booster vaccine uptake at 30 days post ED visit?
* does the intervention of asking about vaccine acceptance increase booster vaccine uptake at 30 days post ED visit?
* considering recent national changes to funding and availability of updated vaccines, the investigators will examine the effects of these changes on vaccine acceptance and uptake in ED populations. Specifically, they will stratify EDs and ED patients according to the ED availability of vaccines, and they will also examine whether costs and availability of vaccines are a deterrent to patient acceptance and uptake of vaccines

DETAILED DESCRIPTION:
I. Overview On January 22, 2020, Acting Health and Human Services Secretary Norris Cochran declared COVID-19 a national public health emergency, an action that eventually enabled emergency authorization for free COVID-19 vaccines, testing and treatments. This public health declaration has been renewed seven times for 90-day intervals, as required under section 319 of the Public Health Service (PHS) Act. Under this declaration over the past two years, the US government has provided full support and distribution of COVID-19 vaccines and therapeutics (antibody therapies, remdesivir, and nirmatrelvir/ritonavir), such that they have been widely available and free of charge to all Americans. Although these measures have not, by any means, ended the pandemic, it is clear from multiple epidemiologic modeling studies that they have decreased hospitalizations and saved hundreds of thousands of lives. They have also led to a narrowing of the profound morbidity and mortality disparities gap that was seen in minority populations in the first two waves of the pandemic.

The PROCOVAXED trial was a multicenter study that sought to decrease COVID-19 vaccine hesitancy and increase COVID-19 vaccine uptake through the use of vaccine messaging platforms in the emergency department (ED). In this trial, investigators found that implementation of our COVID-19 messaging platforms (videos, information sheets and scripted, direct messaging) were associated with greater COVID-19 vaccine acceptance and uptake among unvaccinated ED patients (Rodriguez RM, Nichol G, Eucker SA, et al. Effect of COVID-19 Vaccine Messaging Platforms in Emergency Departments on Vaccine Acceptance and Uptake: A Cluster Randomized Clinical Trial. JAMA Intern Med. 2023;183(2):115-123. doi:10.1001/jamainternmed.2022.5909).

In January 2022, the investigators extended PROCOVAXED by shifting the focus to vaccinated ED patients to examine the timely and critically important topic of booster vaccine hesitancy in underserved ED populations. To better characterize COVID-19 booster hesitancy, the investigators performed a cross-sectional study at five high-volume, safety-net hospital EDs in four cities (San Francisco, Philadelphia, Seattle, and Durham, NC) using survey tools to gather quantitative data on vaccination status, demographic variables, usual source of care, and attitudes toward booster vaccination. Of 771 participants who had completed their full initial series, 316 (41%) had not received any booster vaccine. Among these 316 non-boosted participants, 179 (57%, 95% CI 51-62) stated they would decline or were unsure whether they would accept a booster vaccine if it was offered to them (i.e., booster-hesitant). Investigators found the following associations with booster vaccine hesitancy: age 35-49 years vs age 18-34 years (OR 1.16, 95% CI 0.99-1.36); Asian vs White race (OR 0.21, 95% CI 0.05-0.93); Hispanic/Latino vs White ethnicity (OR 1.59, 95% CI 0.82-3.09); primary language non-English vs English (OR 2.35, 95% CI 1.49-3.71); and Republican vs Democrat party affiliation (OR 6.07, 95% CI 4.21-8.75). The three most common reasons for booster vaccine hesitancy were a preference to wait for more information (25%), concerns about side effects and safety (24%), and "I don't need one because I'm fully vaccinated" (20%).

Recognizing the ED as a unique opportunity to address COVID-19 booster vaccine hesitancy in underserved populations, the investigators will launch the PROmotion of COVID-19 BOOSTer VA(X)ccination in the Emergency Department (PROBOOSTVAXED) trial as an extension of the PROCOVAXED trial, seeking to increase COVID-19 booster vaccine acceptance and uptake among vaccinated ED patients. Because of Omicron variant-associated surges during the COVID-19 pandemic with corresponding research staff illness and ED overcrowding, the investigators found wide week-to-week fluctuations in enrollment in the PROCOVAXED study. To reduce this variability of enrollment, the investigators have changed the unit of randomization from 1-week to 1-day in the PROBOOSTVAXED trial.

As of May 11, 2023, the COVID-19 public health emergency ended. Consequently, not only are the costs for vaccines, testing, and treatments shifted to health insurers and patients via commercial payment mechanisms, but COVID-19 vaccines are no longer available in some EDs. Since our research focuses on the delivery and availability of vaccines to underserved populations whose only health care access occurs in EDs, the team believes that this represents a potential barrier to 30-day vaccine uptake in these populations. The investigators have been informed that only some of the PROBOOSTVAXED study sites will have COVID-19 vaccines available for distribution in the ED, and this availability is subject to change throughout the study period. Nevertheless, the team will proceed with the same research protocol, however, the investigators feel it is important to examine how ED vaccine availability will affect 30-day vaccine uptake in underserved populations. They will therefore be performing additional subgroup analyses that compare 30-day vaccine uptake among sites with available COVID-19 vaccine to those without for the intervention and control arms.They will also evaluate whether patient costs of vaccines are a deterrent to acceptance and uptake.

While the sample size calculation for this research is derived from Aim 1, the investigators emphasize that this is a pragmatic study in which they seek to evaluate the fluid real-world changes in COVID-19 vaccine availability and funding. As stated above, there have been (and likely will continue to be) changes in payment for and availability of vaccines in EDs.

The investigators therefore have developed our protocol and aims below to assess the impact of these changes.

Aim1: To determine whether implementation of COVID-19 booster vaccine trusted messaging platforms is associated with increased booster vaccine uptake in ED patients. At five EDs (Zuckerberg San Francisco General, UCSF Parnassus Medical Center [San Francisco, CA], Thomas Jefferson University Hospital [Philadelphia, PA], Ben Taub Hospital [Houston, TX], Duke University Medical Center [Durham, NC]), investigators will conduct a cluster-randomized controlled trial of the implementation of PROBOOSTVAXED trusted messaging platforms, with 30-day booster vaccine uptake as the primary outcome and booster vaccine uptake in the ED as a secondary outcome. Hypothesis: Implementation of PROBOOSTVAXED trusted messaging platforms in EDs will be associated with increased 30-day booster vaccine uptake in vaccinated ED patients.

Aim 1a: To determine whether implementation of COVID-19 booster vaccine trusted messaging platforms in EDs is associated with increased booster vaccine acceptance in ED patients. For this aim, booster vaccine acceptance in the ED assessed via ED survey will be the primary outcome. Hypothesis: Implementation of PROBOOSTVAXED trusted messaging platforms in EDs will be associated with increased booster vaccine acceptance in ED patients.

Aim 2: To determine whether implementation of a protocol in which ED patients are asked whether they will accept a COVID-19 booster vaccine in the ED is associated with increased booster vaccine uptake in ED patients. Hypothesis: Implementation of an ED protocol in which patients are asked whether they will accept a COVID-19 booster vaccine will be associated with increased 30-day booster vaccine uptake in ED patients.

Aim 3: To compare vaccine uptake (during the index ED visit and 30 days post visit) between sites that have COVID-19 booster vaccine available and those that do not.

Aim 3a: To compare vaccine acceptance and 30-day uptake among patients with health insurance versus those without health insurance (evaluating the effects of patient vaccine cost on acceptance and uptake).

Aim 4: To compare COVID-19 vaccine uptake in this current study with data gathered in our previous COVID-19 vaccine messaging trial.

General Design: This is a three-arm cluster-randomized controlled trial (CRCT).

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Presenting to ED
3. No receipt of COVID-19 booster within prior 6 months
4. Able to provide informed consent
5. Fluent in English or Spanish
6. Anticipated ability to complete study intervention in ED i.e., able to watch a 3-minute videoclip

Exclusion Criteria:

1. Major trauma such that it will preclude survey
2. Inability to participate in a survey because of intoxication, altered mental status, or critical illness
3. Incarceration
4. Psychiatric hold
5. Patients who state that they have already received a bivalent COVID-19 booster vaccine or other COVID-19 vaccine within the prior 6 months
6. Patients who are in the ED for suspected acute COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 919 (Actual)
Dates: Start 2024-01-19 (Actual); Primary Completion 2024-07-18 (Actual); Study Completion 2024-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Rodriguez, MD, Principal Investigator — University of California, San Francisco
Locations (7):
- United States (7):
  - San Francisco General Hospital Emergency Department, San Francisco, California
  - University of California San Francisco Parnassus, San Francisco, California
  - Duke University Hospital, Durham, North Carolina
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Jefferson Torresdale Hospital, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be made available after review of formal request.
Supporting Information: Study Protocol
Time Frame: Upon publication of results
Access Criteria: After review of formal request

REFERENCES:
- [Derived] Molina MF, Eucker SA, Rising KL, Kean ER, Rafique Z, Mesbah H, Glidden DV, Arreguin MI, Alvarez C, Rodriguez RM. COVID-19 Booster Vaccine Messaging in Emergency Departments: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2537655. doi: 10.1001/jamanetworkopen.2025.37655. PMID 41091465

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 919 participants were randomized
Groups:
- Ben Taub Hospital; Duke University Hospital; Jefferson University Hospital: First condition: control
- Jefferson Methodist Hospital; UCSF Parnassus Medical Center; Zuckerberg San Francisco General Hospital: First Condition: Intervention Q
Period: Overall Study
Arm/Group | Ben Taub Hospital | Duke University Hospital | Jefferson University Hospital | Jefferson Methodist Hospital | UCSF Parnassus Medical Center | Zuckerberg San Francisco General Hospital
Started | 132 | 147 | 294 | 3 | 169 | 174
Randomized to Intervention M | 34 | 50 | 84 | 0 | 37 | 63
Randomized to Intervention Q | 52 | 43 | 84 | 1 | 71 | 56
Randomized to Control | 46 | 54 | 126 | 2 | 61 | 55
Completed | 118 | 140 | 279 | 3 | 158 | 154
Not Completed | 14 | 7 | 15 | 0 | 11 | 20
Not completed — Withdrawal by Subject | 2 | 4 | 4 | 0 | 2 | 2
Not completed — Left ED without completing study | 9 | 3 | 9 | 0 | 8 | 16
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Became or found ineligible | 2 | 0 | 2 | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Population: individuals randomized, not withdrawn
Groups:
- PROBOOSTVAXED Intervention M (Messaging + Vaccine Question): * Vaccine messaging
  * Vaccine acceptance question
  Vaccine Messaging: 1) Video clips - short (approximately 3-minute) Public Service Announcement type videos to be viewed by participant using a QR code on their smartphone. If no smartphone is available, the video will be shown to the participant on an iPad.
  2) Printed materials - one page information sheets handed to subjects by CRCs. 3) Face to face messaging - short (< 1 minute), scripted message from the patient's providers in the ED (nurse or provider)
  Each site will maintain a library of
  A. 5 versions of the videos - the version used in any participant will be tailored to that participant's stated race/ethnicity.
  B. 5 versions of printed flyers - likewise, the version will be tailored to the participant's stated race/ethnicity.
  C. 1 version of scripted message to be delivered in English or Spanish.
  Vaccine Acceptance Question: The last question in the Vaccine Acceptance Survey in both the Intervention M and Intervention Q arms of the study is "Would you accept the COVID-19 booster vaccine in the emergency department today if your doctor asked you?"
- Intervention Q (Vaccine Question, No Messaging): * No vaccine messaging
  * Vaccine acceptance question asked in the Vaccine Acceptance Survey
  Vaccine Acceptance Survey: We will administer the Vaccine Acceptance Survey at some time (generally 30 minutes but up to 3 hours) after the Intake Survey. The surveys in the control group retain the same key primary and secondary outcome questions as in the intervention group Vaccine Acceptance surveys.
  Vaccine Acceptance Question: The last question in the Vaccine Acceptance Survey in both the Intervention M and Intervention Q arms of the study is "Would you accept the COVID-19 booster vaccine in the emergency department today if your doctor asked you?"
- Total: Total of all reporting groups
Arm/Group | PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) | Intervention Q (Vaccine Question, No Messaging) | Control (No Messaging, No Vaccine Question) | Total
Number analyzed (Participants) | 247 | 273 | 332 | 852
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [33 to 62] | 49 [33 to 61] | 46 [33 to 61] | 46.5 [33 to 62.5]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Woman | 136 | 142 | 186 | 464
  Man | 107 | 129 | 143 | 379
  Other | 4 | 2 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Participant could identify as more than one race/ethnicity and may be counted in more than one race/ethnicity category
  Participants
    Black | 83 | 85 | 119 | 287
    American Indian, Alaska Native | 3 | 0 | 2 | 5
    Asian | 12 | 20 | 16 | 48
    Latinx | 48 | 61 | 61 | 170
    Middle Eastern | 0 | 0 | 0 | 0
    Native hawaiian/ Pacific Islander | 4 | 4 | 4 | 12
    White (non-Latinx) | 101 | 107 | 137 | 345
    Other | 6 | 8 | 10 | 24
Region of Enrollment [Number; unit: participants]
  United States | 247 | 273 | 332 | 852

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 30-day Booster Vaccine Uptake
Description: Our primary outcome is booster vaccine uptake (at any vaccination location) within 30 days after participants' index ED visit, comparing Intervention M arm with Control
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) | Control (No Messaging, No Vaccine Question)
Number analyzed (Participants) | 247 | 332
Participants | 14 | 10

2. Secondary Outcome: Number or Participants Receiving Booster Vaccination in the ED
Description: Booster vaccine uptake in the ED on the day of the index visit, M arm versus control and Q arm versus control
Time Frame: day of index visit
Measure: Count of Participants; unit: Participants
Arm/Group | PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) | Intervention Q (Vaccine Question, No Messaging) | Control (No Messaging, No Vaccine Question)
Number analyzed (Participants) | 247 | 273 | 332
Participants | 8 | 7 | 0

3. Secondary Outcome: Number of Participants Stating They Would Accept Vaccine in the ED
Description: A response of "yes" to the question, "Would you accept the booster vaccine in the emergency department today if your doctor asked you?"), comparing M and Q arms
Time Frame: on the day of index ED visit
Measure: Count of Participants; unit: Participants
Arm/Group | PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) | Intervention Q (Vaccine Question, No Messaging)
Number analyzed (Participants) | 247 | 273
Participants | 73 | 90

4. Secondary Outcome: Number of Participants With 30-day Booster Vaccine Uptake, Q Arm
Description: Booster vaccine uptake (at any vaccination location) within 30 days after participants' index ED visit, comparing Intervention Q arm with Control
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Q (Vaccine Question, No Messaging) | Control (No Messaging, No Vaccine Question)
Number analyzed (Participants) | 273 | 332
Participants | 11 | 10

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | PROBOOSTVAXED Intervention M (Messaging + Vaccine Question) | Intervention Q (Vaccine Question, No Messaging) | Control (No Messaging, No Vaccine Question)
All-Cause Mortality (participants affected / at risk) | 0/247 | 0/273 | 0/332
Serious Adverse Events (participants affected / at risk) | 0/247 | 0/273 | 0/332
Other Adverse Events (participants affected / at risk) | 0/247 | 0/273 | 0/332

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT06156215/Prot_SAP_000.pdf